CLINICAL TRIAL: NCT01946919
Title: Post-Marketing Surveillance of the Cinepazide Maleate Injection: a Real World Study
Acronym: PACER
Status: Completed | Type: Observational
Sponsor: Peking University Third Hospital (Other)
Collaborators: Beijing Sihuan Pharmaceutical Co. Ltd. (Industry); Beijing Shijitan Hospital,the 9th Clinical Medical College of Peking university (Unknown); China Rehabilitation Research Center (Other Government); Hua Xin Hospital First Hospital of Tsing Hua University (Unknown); Fu Xing Hospital, Capital Medical University (Other); Beijing Chuiyangliu Hospital(Beijing Minimally Invasive Hospital) (Unknown); Dongfang Hospital Beijing University of Chinese Medicine (Other); Dongzhimen Hospital, Beijing (Other); Xuanwu Hospital, Beijing (Other); Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other); Southern Medical University, China (Other); Guangzhou First People's Hospital (Other); Panyu Hospital of Traditional Chinese Medicine (Other); Second Affiliated Hospital of Guangzhou Medical University (Other); The People's Hospital of Gaozhou (Other); Zhongshan Hospital Of Traditional Chinese Medicine (Other); Second Affiliated Hospital of Shantou University Medical College (Other); Sun Yat-sen University (Other); Central People's Hospital of Zhanjiang (Other); Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other); Tongji Hospital (Other); Renmin Hospital of Wuhan University (Other); People's Hospital of Dongxihu District (Unknown); Shenlong Hospital (Unknown); Xiangya Hospital of Central South University (Other); Central South University (Other); The Third Xiangya Hospital of Central South University (Other); Hunan Provincial People's Hospital (Other); The First Affiliated Hospital of Hunan University of Traditional Chinese Medicine (Other); The Third Hospital of Changsha (Unknown); Ankang City Central Hospital (Other); San Er Ling Yi Hospital (Unknown); Xijing Hospital (Other); Tang-Du Hospital (Other); First Affiliated Hospital Xi'an Jiaotong University (Other); Gansu Provincial Hospital (Other); Xi'an Central Hospital (Other); LanZhou University (Other); Qilu Hospital of Shandong University (Other); Binzhou People's Hospital (Other); Jiangxi Provincial People's Hopital (Other); The First Affiliated Hospital of Nanchang University (Other); Second Affiliated Hospital of Nanchang University (Other); The Third Affiliated Hospital of Nanchang University (Other); The Third Hospital of Nanchang (Unknown); First Affiliated Hospital of Harbin Medical University (Other); First Affiliated Hospital of Heilongjiang Chinese Medicine University (Other); People's Hospital of Heilongjiang Province (Unknown); The Second Affiliated Hospital of Harbin Medical University (Other); The first hospital of Harbin City (Unknown); The Fourth Affiliated Hospital of Harbin Medical University (Other); Second Affiliated Hospital of Heilongjiang University of Chinese Medicine (Other); First Hospital of China Medical University (Other); People's Liberation Army No.202 Hospital (Other); The Fourth Affiliated Hospital of China Medical University (Other); General Hospital of Shenyang Military Region (Other); The four six three hospital of people's Liberation Army (Unknown); First People's Hospital of Shenyang (Other); Jilin Province People's Hospital (Unknown); Beihua University (Other); Shenzhou Hospital to Shenyang Medical College (Unknown)
Responsible Party: Principal Investigator, Suodi ZHAI, Suodi ZHAI, Department of Pharmacy, Peking University Third Hospital, Peking University Third Hospital
Other Study IDs: PekingUTH-Pharmacy-002
Record Dates: First submitted 2013-09-12; First posted 2013-09-20 (Estimated); Last update posted 2022-07-27 (Actual); Status verified 2022-07

CONDITIONS: Adverse Drug Reaction; Cinepazide; Stroke
Keywords: Cinepazide; Adverse Drug Reaction; Safety; Real World Study
MeSH Terms: conditions — Drug-Related Side Effects and Adverse Reactions; Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 14 Days
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- cinepazide: Inpatient using the cinepazide in department of neurology

SUMMARY:
Cinepazide Maleate Injection is widely used in cerebrovascular disease in china. The safety of the cinepazide, especially the blood system, has not been fully evaluated in Chinese population. In order to improve the rational use of cinepazide, the investigators observe its clinical use in the real world in China, evaluate its safety and clinical benefit in a large Chinese population.

DETAILED DESCRIPTION:
Cinepazide was firstly approved in France in 1974, and the formulations are injection and tablet. Products containing cinepazide have been withdrawn in 1990s by the manufacturers because of lacking of demonstrated efficacy and the risk of agranulocytosis in some European countries, such as France, Spain, Italy. In some Aisa countries, it has not been re-registered in Japan in 2000s, and the injection is still used in China and Korea. In china, Cinepazide Maleate Injection was approved by China Food and Drug Administration(CFDA) in 2002, and widely used in cerebrovascular disease. The safety of the Cinepazide, especially the adverse drug reactions in the blood system, has not benn fully evaluated in Chinese population. In this study, clinical pharmacists in selected hospitals will record the clinical use and the adverse drug reactions/ adverse drug events of this injection. This real world study for Cinepazide Maleate Injection with 18000 patients will be conducted from Sep. 2012 to June. 2014.

ELIGIBILITY:
Inclusion Criteria:

* Inpatient using the cinepazide in the department of neurology

Exclusion Criteria:

* none

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Inpatient using the cinepazide in the department of neurology in 61 hospitals in China.
Sampling Method: Non-Probability Sample
Enrollment: 18260 (Actual)
Dates: Start 2012-10; Primary Completion 2021-12 (Actual); Study Completion 2022-06 (Actual)

PRIMARY OUTCOMES:
Incidence of adverse drug reaction of cinepazide in department of neurology | 1.5 years

SECONDARY OUTCOMES:
Outcomes of the patients who experienced an adverse drug reaction of cinepazide. | 1.5 years
  Outcomes including cure, improved, null, or death.
The predictors of the adverse drug reaction of cinepazide | 1.5 years
  We will analyse whether some factors, such as age, gender, medical history and etc, would be the predictors of the adverse drug reaction of cinepazide.
Types of the adverse drug reaction of cinepazide. | 1.5 years
  The types of the adverse drug reaction of cinepazide including Nausea, vomiting, itching and etc.
The treatment when patients experienced an adverse drug reaction of cinepazide. | 1.5 years
  Treatments including oxygen, steroids, and etc. According to severity of the adverse drug reactions, we will analyse the features the treatments, such as types and numbers.

CONTACTS AND LOCATIONS:
Locations (61):
- China (61):
  - China Rehabilitation Research Center, Beijing, Beijing Municipality
  - Dongfang Hospital,the second clinical medical College of Beijing University of Chinese Medicine(BUCM), Beijing, Beijing Municipality
  - Dongzhimen Hospital Affiliated to Beijing University of Chinese Medicine, Beijing, Beijing Municipality
  - Fu Xing Hospital,Capital Medical University, Beijing, Beijing Municipality
  - Beijing Chuiyangliu Hospital(Beijing Minimally Invasive Hospital), Beijing, Beijing Municipality
  - Hua Xin Hospital; First Hospital of Tsing Hua University, Beijing, Beijing Municipality
  - Xuanwu Hospital Affiliated to Capital Medical University, Beijing, Beijing Municipality
  - Beijing Shijitan Hospital,the 9th Clinical Medical College of Peking university, Beijing, Beijing Municipality
  - Peking University Third Hospital, Beijing, Beijing Municipality
  - Gansu Provincial Hospital, Lanzhou, Gansu
  - The First Affiliated Hospital of Lanzhou University, Lanzhou, Gansu
  - Central People's Hospital of Zhanjiang, Ganjiang, Guangdong
  - The People's Hospital of Gaozhou, Gaozhou, Guangdong
  - GuangZhou First People's Hospital, Guangzhou, Guangdong
  - Panyu Hospital of Chinese Medicine, Guangzhou, Guangdong
  - Sun Yat-Sen Memorial Hospital Sun Yat-Sen University, Guangzhou, Guangdong
  - The Second Affiliated Hospital of Guangzhou Medical University, Guangzhou, Guangdong
  - ZhuJiang Hospital of Southern Medical University, Guangzhou, Guangdong
  - Shantou Central Hospital Affiliated Shantou Hospital of Sun Yan-Sen University, Shantou, Guangdong
  - The Second Affiliated Hospital of Shantou University Medical College, Shantou, Guangdong
  - Hospital of Traditional Chinese Medicine of Zhongshan, Zhongshan, Guangdong
  - People's Hospital of Dongxihu District, Wuhan, Hebei
  - Shenlong Hospital, Wuhan, Hebei
  - People's Hospital of Heilongjiang Province, Harbin, Heilongjiang
  - The 2nd Affiliated Hospital of Harbin Medical University, Harbin, Heilongjiang
  - The First Affiliated Hospital of Harbin Medical University, Harbin, Heilongjiang
  - The First Affiliated Hospital of Heilongjiang University Of Chinese Medicine, Harbin, Heilongjiang
  - The first hospital of Harbin City, Harbin, Heilongjiang
  - The Fourth Affiliated Hospital of Harbin Medical University, Harbin, Heilongjiang
  - The Second Affiliated of Heilongjiang University of Chinese Medicine, Harbin, Heilongjiang
  - Renmin Hospital of Wuhan, Wuhan, Hubei
  - Tongji Hospital, Wuhan, Hubei
  - Wuhan Union Hospital, Wuhan, Hubei
  - Hunan Provincial People's Hospital, Changsha, Hunan
  - The First Hospital of Changsha, Changsha, Hunan
  - The Second Xiangya Hospital of Central South University, Changsha, Hunan
  - The Third Hospital of Changsha, Changsha, Hunan
  - The Third Xiangya Hospital of Central South University, Changsha, Hunan
  - Xiangya Hospital Central-South University, Changsha, Hunan
  - Jiangxi Provincial People's Hospital, Nanchang, Jiangxi
  - The First Affiliated Hospital of Nanchang University, Nanchang, Jiangxi
  - The Second Affiliated Hospital of Nanchang University, Nanchang, Jiangxi
  - The Third Affiliated Hospital of Nanchang University, Nanchang, Jiangxi
  - The Third Hospital of Nanchang, Nanchang, Jiangxi
  - Jilin Province People's Hospital, Changchun, Jilin
  - Affiliated Hospital of Beihua University, Jilin, Jilin
  - General Hospital of Shenyang military area command of Chinese PLA, Shenyang, Liaoning
  - Shenyang First People's Hospital, Shenyang, Liaoning
  - Shenzhou Hospital to Shenyang Medical College, Shenyang, Liaoning
  - The First Affiliated Hospital of China Medical University, Shenyang, Liaoning
  - The four six three hospital of people's Liberation Army, Shenyang, Liaoning
  - The Fourth Affiliated Hospital of China Medical University, Shenyang, Liaoning
  - The people's Liberation Army 202nd hospital, Shenyang, Liaoning
  - Ankang City Central Hospital, Ankang, Shaanxi
  - San Er Ling Yi Hospital, Hanzhong, Shaanxi
  - First Affiliated Hospital of Medical College of Xian Jiaotong University, Xi'an, Shaanxi
  - Tangdu Hospital, Xi'an, Shaanxi
  - The Central Hospital of Xi'an, Xi'an, Shaanxi
  - Xijing Hospital, Xi'an, Shaanxi
  - Binzhou People's Hospital, Binzhou, Shandong
  - Qilu Hospital of Shandong University, Jinan, Shandong